CLINICAL TRIAL: NCT03638245
Title: Evaluation of the Fetal Myocardial Performance Index in Abnormal Cardiotocography Cases in 3rd Trimester of Pregnancy and Fetal Outcome
Brief Title: Evaluation of the Fetal MPI in Abnormal Cardiotocography Cases in 3rd Trimester of Pregnancy and Fetal Outcome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ali Mohamed AbdEl-Halim Ali Mehanna (Other)
Responsible Party: Sponsor-Investigator, Ali Mohamed AbdEl-Halim Ali Mehanna, Dr, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: USCU 230
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal CTG: This group includes pregnancies that showed abnormalities in CTG.
- Normal CTG: This group includes pregnancies that showed no abnormalities in CTG.

SUMMARY:
The study will focus in evaluation of fetal cardiac function by using myocardial performance index in fetuses with abnormal cardiotocography in 3rd trimester.

DETAILED DESCRIPTION:
The study will focus in evaluation of fetal cardiac function by using myocardial performance index in fetuses with abnormal cardiotocography in 3rd trimester.

Study Hypothesis:

In women with non reassuring fetal cardiotocography, myocardial performance index may predict fetal distress accurately.

Study Question:

In pregnant women in the third trimester with abnormal cardiotocography, Does myocardial performance index predict fetal distress accurately?

Study Objectives:

This study aims to assess the accuracy of myocardial performance index in predicting fetal distress in pregnant women with non reassuring cardiotocography in third trimester.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 30-40 weeks gestational age.
2. Women pregnant in singleton fetus.

Exclusion Criteria:

1. Multiple pregnancies.
2. Fetal congenital malformation.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women in 3rd trimester attending for CTG
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2019-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Fetal Myocardial Performance Index. | 3rd Trimester CTG, immediately followed by Fetal Echocardiography at the same set
  Evaluation of the Fetal Myocardial Performance Index in Abnormal Cardiotocography Cases in 3rd Trimester of Pregnancy and Fetal Outcome.

SECONDARY OUTCOMES:
Neonatal outcome observation | Immediately postnatal (first five minutes after delivery)
  APGAR score at the first and fifth minute

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Nasr El din, MD, Study Chair — Professor; Amr MA El Helaly, MD, Study Director — Assistant Professor; Noha AA Sakna, MD, Study Director — Lecturer